CLINICAL TRIAL: NCT04466189
Title: Prospective Cohort Study for Identifying Factors Predicting Clinical Outcomes of Pancreatic Cancer Patients Treated With Proton Beam Therapy
Brief Title: Prospective Cohort Study of Pancreatic Cancer Patients Treated With Proton Beam Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Tae Hyun Kim, Principal Investigator, National Cancer Center, Korea
Other Study IDs: NCC2018-0198
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Pancreas Cancer
Keywords: Proton Beam Therapy; Cohort Study
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatic Cancer Patients Treated With Proton Beam Therapy: Pancreatic Cancer Patients Treated With Proton Beam Therapy

SUMMARY:
Pancreatic cancer is one of the few cancers whose survival rate has not improved significantly due to high local recurrence and systemic metastasis despite advances in diagnosis and treatment over the past 40 years. And currently pancreatic cancer is the fifth leading cause of cancer-related death in Korea. For this reason, various anti-cancer therapies and radiotherapy have been tested to improve survival.

Due to recent advances in radiotherapy technology, proton beam therapy (PBT) is a promising treatment for pancreatic cancer because it can reduce radiation dose from surrounding normal tissue while maximizing radiation to tumor tissues due to the distinct physical properties of proton beam. Low toxicity have been reported. In addition, retrospective analysis of pancreatic cancer patients (n=37) who performed proton therapy (PBT) from June 2013 to July 2016 showed promising therapeutic performance and less toxicity (survival rate, 19.3 months; Grade ≥ 3 Toxicity, 0%). In addition, gene polymorphisms of several genes (CD44, CD166, XAF1, MMP9, MUC1/4, SMAD7, SMAD4 (DPC), RRM1, ERCC1, HER2, etc.) in pancreatic cancer have been reported to be associated with recurrence and prognosis.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the few cancers whose survival rate has not improved significantly due to high local recurrence and systemic metastasis despite advances in diagnosis and treatment over the past 40 years. And currently pancreatic cancer is the fifth leading cause of cancer-related death in Korea. For this reason, various anti-cancer therapies and radiotherapy have been tested to improve survival.

Due to recent advances in radiotherapy technology, proton beam therapy (PBT) is a promising treatment for pancreatic cancer because it can reduce radiation dose from surrounding normal tissue while maximizing radiation to tumor tissues due to the distinct physical properties of proton beam. Low toxicity have been reported. In addition, retrospective analysis of pancreatic cancer patients (n=37) who performed proton therapy (PBT) from June 2013 to July 2016 showed promising therapeutic performance and less toxicity (survival rate, 19.3 months; Grade ≥ 3 Toxicity, 0%). In addition, gene polymorphisms of several genes (CD44, CD166, XAF1, MMP9, MUC1/4, SMAD7, SMAD4 (DPC), RRM1, ERCC1, HER2, etc.) in pancreatic cancer have been reported to be associated with recurrence and prognosis. Therefore, in this study, a prospective cohort of pancreatic cancer patients treated with proton beam therapy was established to analyze local control, survival, recurrence, toxicity, proton treatment plan information, gene expression information to analyze local control (LC), overall survival (OS), recurrence-free surival (RFS), and factors predicting treatment-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer patients scheduled to be proton beam therapy
* Agreed to participate in this study

Exclusion Criteria:

-Disagreed to participate in this study

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients over the age of 19
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Establish a cohort of Pancreatic cancer patients treadted with proton beam therapy. | Up to 10 years
  The primary outcome is to establish a prospective cohort of pancreatic cancer patients treadted with proton beam therapy. It is for exploring factors and models that predict local control, relapse, survival and treatment-related toxicity in patients with pancreatic cancer who have undergone proton therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Hyun Kim, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea